CLINICAL TRIAL: NCT00827411
Title: Double Randomization of a Monitoring Adjusted Antiplatelet Treatment Versus a Common Antiplatelet Treatment for DES Implantation, and a Interruption Versus Continuation of Double Antiplatelet Therapy, One Year After Stenting
Brief Title: Double Randomization of a Monitoring Adjusted Antiplatelet Treatment Versus a Common Antiplatelet Treatment for DES Implantation, and Interruption Versus Continuation of Double Antiplatelet Therapy
Acronym: ARCTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Allies in Cardiovascular Trials Initiatives and Organized (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Sanofi (Industry); Bristol-Myers Squibb (Industry); Medtronic (Industry); Cordis US Corp. (Industry); Fondation de France (Other); Diagnostica Stago (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080403
Record Dates: First submitted 2009-01-13; First posted 2009-01-22 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Drug Eluting Stent; Percutaneous coronary intervention; Oral antiplatelet therapy; Clopidogrel/Aspirin; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Monitoring Arm (Experimental): First randomization:
  Monitoring Arm: dose adjustment of both aspirin and clopidogrel in suboptimal responders identified based on a point of care assay (VerifyNow).
  Interventions: Drug: Aspirin and clopidogrel / Prasugrel; Device: VerifyNow
- 2: Conventional Arm (Active Comparator): First randomization:
  Conventional Arm: fixed dose regiment of both aspirin and clopidogrel in all patients following DES implantation according to international guidelines
  Interventions: Drug: Aspirin and clopidogrel / Prasugrel
- 3: Pursuit Arm (Experimental): Second randomization after one year of follow-up:
  Pursuit Arm: Pursuit of a dual oral antiplatelet therapy (aspirin and clopidogrel) beyond one year
  Interventions: Drug: Aspirin and clopidogrel / Prasugrel
- 4: Interruption Arm (Active Comparator): Second randomization after one year of follow-up:
  Interruption Arm: Interruption of clopidogrel therapy.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin and clopidogrel / Prasugrel — modification of aspirin and clopidogrel/Prasugrel maintenance doses based on a biological assay
  Arms: 1: Monitoring Arm
Device: VerifyNow — point of care assay VerifyNow (ACCUMETRICS San Diego USA)
  Arms: 1: Monitoring Arm
Drug: Aspirin and clopidogrel / Prasugrel — aspirin and clopidogrel/ Prasugrel maintenance doses (according to international guidelines)
  Arms: 2: Conventional Arm
Drug: Aspirin and clopidogrel / Prasugrel — maintenance dose of clopidogrel / Prasugrel and aspirin
  Arms: 3: Pursuit Arm
Drug: Aspirin — Interruption of clopidogrel / Prasugrel after one year of follow-up
  Arms: 4: Interruption Arm

SUMMARY:
Our first hypothesis is that dose adjustment of aspirin and clopidogrel based on biological monitoring reduces the rate of severe cardiovascular complications compared to a conventional strategy in patients scheduled for drug eluting stent implantation and followed up for one year. Our second hypothesis is that interruption of clopidogrel / Prasugrel after one year of a combined therapy of clopidogrel/Prasugrel and aspirin is associated with a higher rate of severe cardiovascular complications as compared with patients in whom aspirin and clopidogrel / Prasugrel is maintained during the subsequent 6 months of follow-up.

DETAILED DESCRIPTION:
Participating Centers : 38 french high PCI volume (>700) centers Rationale: Clopidogrel / Prasugrel (75 mg/day), in combination with aspirin (75 mg/day), is currently the antiplatelet treatment of choice for prevention of stent thrombosis, and clinical trials have shown that, in high-risk patients, prolonged dual antiplatelet treatment is more effective than aspirin alone in preventing major cardiovascular events. However, despite the use of clopidogrel, a considerable number of patients continue to have cardiovascular events. Numerous in VITRO studies have shown that individual responsiveness to clopidogrel but also to aspirin is not uniform in all patients and is subject to inter- and intraindividual variability. The recent possibility of bedside monitoring of oral antiplatelet therapy offers the unique opportunity of tailoring antiplatelet therapy. However, the relevance of such strategy has never been evaluated in a randomized prospective adequately powered study having long term follow-up (rationale 1). Late state stent thrombosis, especially in the era of drug eluting stent and after interruption of OAT, is another important safety issue raising the questions of the modalities of interruption of dual OAT after one year according to the most recent updated recommendations. Can we switch from dual to single OAT after one year? If so, what is the ischemic hazard? (Rational 2) Our first hypothesis is that a strategy of dose adjustment of OAT based on biological monitoring reduces the rate of the combined ischemic endpoints of death, urgent revascularization, stent thrombosis and stroke as compared to a conventional strategy (local practice without monitoring) in patients scheduled for DES implantation and followed up for one year. Our second hypothesis is that interruption of clopidogrel after one year of dual OAT is associated with a higher rate of the same combined ischemic endpoints as compared with patients in whom dual OAT is maintained during the subsequent 6 months of follow-up. Objectives: 1) To demonstrate the superiority of the strategy of monitoring with dose adjustment in suboptimal responders (Monitoring Arm) as compared to a more conventional strategy (Conventional Arm) with fixed dose regimen of both oral antiplatelet agents in all patients as defined by the international guidelines to reduce the primary endpoint evaluated one year after DES implantation. 2) to demonstrate the superiority of a strategy of pursuit of a dual OAT beyond one year (Pursuit Arm) as compared to a strategy of interruption (Interruption Arm).

Duration of the participation : from 18 up to 30 months according to the time delay from study start to randomization. No participants will be excluded from the study at the exception of consent withdrawal. However, participants who have not been randomized for interruption or continuation of DAPT at the 12 month follow up visit will terminate the study

Number of patients: 2500 patients. This number was obtained for the demonstration of the superiority of the strategy of monitoring (Monitoring Arm) over the conventional strategy (Conventional Arm) to reduce the primary endpoint by 33% (relative risk reduction).

Expected results: The ARCTIC study will provide answers to two major clinical challenges. It will also give a unique opportunity to assess the prevalence and the associated risk factors of suboptimal answers to OAT, but also to improve a suboptimal biological response. Finally, the economic impact of both strategies of monitoring and of interruption will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years) in whom elective DES stent placement is scheduled after diagnostic angiography
* Patients not treated by GPIIb/IIIa inhibitors prior to randomization.
* Provided written consent for participation in the trial prior to any study-specific procedures or requirements.

Exclusion Criteria:

* Oral anticoagulation (Vitamin K Antagonists).
* Contraindication for aspirin and/or clopidogrel/Prasugrel or GPIIb/IIIa inhibitors or to increasing dose of clopidogrel or aspirin
* Ongoing or recent bleeding and/or recent major surgery (<3 weeks)
* Severe liver dysfunction
* Thrombocytopenia (Platelet count <80000/µl).
* IIb/IIIa inhibitors within a week prior to randomization
* STEMI presentation
* Patient at risk of poor compliance to the study
* Patient not affiliated to social security
* Pregnant women, no signed inform consent
* Any invasive or surgical planned intervention during the year after stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of death, myocardial infarction, stroke, urgent coronary revascularization, stent thrombosis assessed at one year for the first hypothesis and between 6 up to 18 months of follow-up for the second hypothesis | during the study (one year in both " monitoring " and " conventional " arms and during the periode from 6 up to 18 months in the "interruption" and "pursuit" arms)

SECONDARY OUTCOMES:
Stent thrombosis and urgent coronary revascularization | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Rate of individual event at one year follow-up in both " monitoring " and " conventional " arms but also during the period from one year up to 24 months in the " interruption " and " pursuit " arms. | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Time delay from treatment interruption (randomization 2) to any thrombotic event (stent thrombosis, urgent revascularization, acute myocardial infarction, cardiac death) treatment interruption(randomisation 2) | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Treatment compliance evaluated by the number of oral antiplatelet treatment in both arms and with respect to all individual events of the primary composite endpoint | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Rate of use of GP IIb/IIIa receptor antagonists in both " monitoring " and " conventional " arms before percutaneous coronary intervention and in bail out situations and in both. | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Rate of suboptimal responders as defined by ARU>550 for aspirin or by a % of inhibition <15% and or a PRU<235) and the average dosage of aspirin and clopidogrel (in mg) will evaluated before and after dose adjustment (J0) and after each dose adjustment | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Net clinical benefit (death, myocardial infarction, urgent revascularization, stent thrombosis, stroke, major bleeding) | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient
Medico-economic evaluations will be performed for both hypotheses. The rate of rehospitalisation and the length of stay will be used as economic indicators | at month 12 and month 30
  * at month 12 for the non-randomized patients at M12
  * at month 12 and month 30 for the randomized patient

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Montalescot, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris; Jean-Philippe Collet, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Institut de Cardiologie- Hopital la Pitié Salpétrière, Paris, France

REFERENCES:
- [Result] Collet JP, Cuisset T, Range G, Cayla G, Elhadad S, Pouillot C, Henry P, Motreff P, Carrie D, Boueri Z, Belle L, Van Belle E, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Barthelemy O, Beygui F, Silvain J, Vicaut E, Montalescot G; ARCTIC Investigators. Bedside monitoring to adjust antiplatelet therapy for coronary stenting. N Engl J Med. 2012 Nov 29;367(22):2100-9. doi: 10.1056/NEJMoa1209979. Epub 2012 Nov 4. PMID 23121439
- [Result] Collet JP, Cayla G, Cuisset T, Elhadad S, Range G, Vicaut E, Montalescot G. Randomized comparison of platelet function monitoring to adjust antiplatelet therapy versus standard of care: rationale and design of the assessment with a double randomization of (1) a fixed dose versus a monitoring-guided dose of aspirin and clopidogrel after DES implantation, and (2) treatment interruption versus continuation, 1 year after stenting (ARCTIC) study. Am Heart J. 2011 Jan;161(1):5-12.e5. doi: 10.1016/j.ahj.2010.09.029. PMID 21167334
- [Derived] Lattuca B, Silvain J, Yan Y, Pouillot C, Cuisset T, Cayla G, Henry P, Diallo A, Elhadad S, Range G, Lhermusier T, Boueri Z, Motreff P, Carrie D, Vicaut E, Montalescot G, Collet JP. Reasons for the Failure of Platelet Function Testing to Adjust Antiplatelet Therapy: Pharmacodynamic Insights From the ARCTIC Study. Circ Cardiovasc Interv. 2019 Nov;12(11):e007749. doi: 10.1161/CIRCINTERVENTIONS.118.007749. Epub 2019 Nov 7. PMID 31694410
- [Derived] Collet JP, Hulot JS, Cuisset T, Range G, Cayla G, Van Belle E, Elhadad S, Rousseau H, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Barthelemy O, Beygui F, Silvain J, Vicaut E, Montalescot G; ARCTIC investigators. Genetic and platelet function testing of antiplatelet therapy for percutaneous coronary intervention: the ARCTIC-GENE study. Eur J Clin Pharmacol. 2015 Nov;71(11):1315-24. doi: 10.1007/s00228-015-1917-9. Epub 2015 Aug 13. PMID 26265231
- [Derived] Collet JP, Silvain J, Barthelemy O, Range G, Cayla G, Van Belle E, Cuisset T, Elhadad S, Schiele F, Lhoest N, Ohlmann P, Carrie D, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Beygui F, Vicaut E, Montalescot G; ARCTIC investigators. Dual-antiplatelet treatment beyond 1 year after drug-eluting stent implantation (ARCTIC-Interruption): a randomised trial. Lancet. 2014 Nov 1;384(9954):1577-85. doi: 10.1016/S0140-6736(14)60612-7. Epub 2014 Jul 15. PMID 25037988
- [Derived] Montalescot G, Range G, Silvain J, Bonnet JL, Boueri Z, Barthelemy O, Cayla G, Belle L, Van Belle E, Cuisset T, Elhadad S, Pouillot C, Henry P, Motreff P, Carrie D, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Beygui F, Vicaut E, Collet JP; ARCTIC Investigators. High on-treatment platelet reactivity as a risk factor for secondary prevention after coronary stent revascularization: A landmark analysis of the ARCTIC study. Circulation. 2014 May 27;129(21):2136-43. doi: 10.1161/CIRCULATIONAHA.113.007524. Epub 2014 Apr 9. PMID 24718568